CLINICAL TRIAL: NCT07221084
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Assess Pharmacokinetics, Safety, and Tolerability of Atumelnant in Healthy Japanese and Caucasian Participants
Brief Title: A Study to Assess Pharmacokinetics, Safety, and Tolerability of Atumelnant in Healthy Japanese and Caucasian Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRN04894-153
Record Dates: First submitted 2025-10-22; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; CRN04894; Atumelnant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment (Cohort 1) (Experimental): Fixed-sequence cohort for Japanese participants.
  Interventions: Drug: Atumelnant
- Placebo (Cohort 1) (Active Comparator): Fixed-sequence cohort for Japanese participants.
  Interventions: Drug: Placebo
- Treatment (Cohort 2) (Experimental): Fixed-sequence cohort for Caucasian participants.
  Interventions: Drug: Atumelnant
- Placebo (Cohort 2) (Active Comparator): Fixed-sequence cohort for Caucasian participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atumelnant — Atumelnant, tablets, once daily by mouth
  Other Names: CRN04894
  Arms: Treatment (Cohort 1); Treatment (Cohort 2)
Drug: Placebo — Placebo, tablets, once daily by mouth
  Arms: Placebo (Cohort 1); Placebo (Cohort 2)

SUMMARY:
The purpose of this study is to assess the PK profile, safety, and tolerability of atumelnant after single and multiple once daily (QD) oral doses in healthy Japanese and Caucasian adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, stratified randomized, double-blind, placebo-controlled, 2-cohort, 2-period, fixed-sequence study to assess the PK profile, safety, and tolerability of atumelnant after single and multiple QD oral doses in healthy Japanese and Caucasian adult participants.

Approximately 20 healthy male and female participants of either Japanese or Caucasian ethnicities will be enrolled in the study to receive the study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants, 18 to 55 years old, inclusive, at the Screening Visit.
* Healthy status as defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, clinical chemistry, coagulation, serology, and urinalysis. The tests may be repeated once at Screening and at admission on Day -1 if necessary and deemed appropriate by the Investigator or designee.
* Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at the Screening Visit and at admission on Day -1.
* Meeting the criteria at the time of consent for one of the following ethnic groups:
* Japanese participants must have been born in Japan to parents and grandparents of Japanese ethnic descent as evidenced by verbal confirmation and documented in a self-reported family tree form, have lived less than 10 years outside of Japan, and have no significant change in lifestyle, including diet, since leaving Japan.
* Caucasian participants must be considered White of European descent.
* Participant has a peak 30- or 60-minute ACTH stimulated serum cortisol ≥18 μg/dL during 250 μg high-dose ACTH/cosyntropin stimulation test conducted at Screening.
* Participant has normal morning serum cortisol collected at approximately 08:00 AM (±2 hours) at admission on Day -1 and does not have signs and symptoms of adrenal insufficiency as deemed by the Investigator or designee.

Exclusion Criteria:

* Participant is breastfeeding or has a positive serum pregnancy test at Screening or at admission on Day -1.
* Participant has a blood loss ≥500 mL or donated blood within 3 months prior to admission on Day -1.
* Participant has received atumelnant previously or has previously been enrolled in this clinical study.
* Participant has received any investigational drug within the past 30 days or 5 half lives, whichever is longer, prior to the first dose of study intervention on Day 1.
* Participant is unwilling to refrain from strenuous, unaccustomed exercise and sports, defined as greater than 30 minutes per day, 3 days prior to admission on Day -1.
* Participant has history of hypersensitivity to study intervention or any of the excipients or to medicinal products with similar chemical structures.
* Participant has used any prescription medication without approval of the Investigator or designee within 14 days prior to admission on Day -1. By exception, hormonal contraceptives are permitted throughout the study and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines are allowed up to 14 days prior to admission on Day -1.
* Venous access considered inadequate for sample collection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax) | [Time Frame: Up to Day 30]
  Assessment of the maximum observed plasma concentration of atumelnant
Pharmacokinetics (Tmax) | [Time Frame: Up to Day 30]
  Assessment of time to maximal atumelnant concentration (Tmax)
Pharmacokinetics (AUC) | [Time Frame: Up to Day 30]
  Assessment of the plasma area under the curve of Atumelnant

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events including Adverse Events of Special Interest (adrenal insufficiency) | [Time Frame: Up to Day 50]
Number of participants with clinically significant clinical laboratory abnormalities | [Time Frame: Up to Day 30]
Number of participants with clinically significant changes in vital signs | [Time Frame: Up to Day 30]
Number of participants with clinically significant changes in physical exam observations | [Time Frame: Up to Day 30]
Number of participants with clinically significant Electrocardiogram (ECG) abnormalities | [Time Frame: Up to Day 20]
12-lead triplicate Electrocardiogram (ECG) corrected QT interval (QTc) interval | [Time Frame: Up to Day 20]

CONTACTS AND LOCATIONS:
Locations (1):
- Crinetics Study Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No